CLINICAL TRIAL: NCT05287256
Title: Comparative Pharmacokinetic and Pharmacodynamic Effects of Delta-8 and Delta-9 THC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Substance Abuse and Mental Health Services Administration (SAMHSA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB00321661
Record Dates: First submitted 2022-03-10; First posted 2022-03-18 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Behavioral Pharmacology of Cannabis
MeSH Terms: interventions — nabiximols

STUDY DESIGN:
Intervention Model Description: A within-subjects design. At the time of study randomization, participants will be assigned to complete Sub-Study 1 followed by Sub-Study 2, or vice versa, using a counter-balanced randomization sequence. The order in which dose conditions are administered within each sub-study will be randomized across participants because there are too many drug conditions to fully counterbalance dosing within sub-studies at the proposed sample size.
Who Masked: Participant, Care Provider
Masking Description: Placebo controlled, double blind drug administration
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Placebo Oral Cannabis (Placebo Comparator): Single acute administration of placebo cannabis baked into a brownie
  Interventions: Drug: Oral Placebo
- Oral administration of 10mg D-8-THC (Experimental): Single acute administration of cannabis containing 10mg Delta-8-THC baked into a brownie
  Interventions: Drug: Oral Delta-8-THC Cannabis
- Oral administration of 20mg D-8-THC (Experimental): Single acute administration of cannabis containing 20mg Delta-8-THC baked into a brownie
  Interventions: Drug: Oral Delta-8-THC Cannabis
- Oral administration of 40mg D-8-THC (Experimental): Single acute administration of cannabis containing 40mg Delta-8-THC baked into a brownie
  Interventions: Drug: Oral Delta-8-THC Cannabis
- Oral administration of 20mg D-9-THC (Experimental): Single acute administration of cannabis containing 20mg Delta-9-THC baked into a brownie
  Interventions: Drug: Oral Delta-9-THC Cannabis
- Placebo Vaporized Cannabis (Placebo Comparator): Single acute administration of placebo cannabis via commercial vaporizer
  Interventions: Drug: Vaporized Placebo
- Administration of vaporized 10mg D-8-THC (Experimental): Single acute administration of placebo cannabis containing 10mg Delta-8-THC via commercial vaporizer
  Interventions: Drug: Vaporized Delta-8-THC Cannabis
- Administration of vaporized 20mg D-8-THC (Experimental): Single acute administration of placebo cannabis containing 20mg Delta-8-THC via commercial vaporizer
  Interventions: Drug: Vaporized Delta-8-THC Cannabis
- Administration of vaporized 40mg D-8-THC (Experimental): Single acute administration of placebo cannabis containing 40mg Delta-8-THC via commercial vaporizer
  Interventions: Drug: Vaporized Delta-8-THC Cannabis
- Administration of vaporized 20mg D-9-THC (Experimental): Single acute administration of placebo cannabis containing 20mg Delta-9-THC via commercial vaporizer
  Interventions: Drug: Vaporized Delta-9-THC Cannabis

INTERVENTIONS:
Drug: Oral Delta-8-THC Cannabis — Delta-8-THC cannabis will be orally self-administered by study participants
  Other Names: marijuana
  Arms: Oral administration of 10mg D-8-THC; Oral administration of 20mg D-8-THC; Oral administration of 40mg D-8-THC
Drug: Oral Delta-9-THC Cannabis — Delta-9-THC cannabis will be orally self-administered by study participants
  Other Names: marijuana
  Arms: Oral administration of 20mg D-9-THC
Drug: Oral Placebo — Placebo will be orally self-administered by study participants
  Arms: Placebo Oral Cannabis
Drug: Vaporized Delta-8-THC Cannabis — Delta-8-THC cannabis will be self-administered by study participants using a vaporizer
  Other Names: marijuana
  Arms: Administration of vaporized 10mg D-8-THC; Administration of vaporized 20mg D-8-THC; Administration of vaporized 40mg D-8-THC
Drug: Vaporized Delta-9-THC Cannabis — Delta-9-THC cannabis will be self-administered by study participants using a vaporizer
  Other Names: marijuana
  Arms: Administration of vaporized 20mg D-9-THC
Drug: Vaporized Placebo — Placebo will be self-administered by study participants using a vaporizer
  Arms: Placebo Vaporized Cannabis

SUMMARY:
The current study will investigate the subjective, physiological, and cognitive performance effects of inhaled and orally ingested Delta-8 tetrahydrocannabinol (THC) in comparison to both placebo and Delta-9 THC. The purpose of this study is to assess the effects of Delta-8 THC as compared to placebo and Delta-9 THC. Oral fluid, urine, blood, and hair specimens will be collected from participants.

DETAILED DESCRIPTION:
The current study will investigate the subjective, physiological, and cognitive performance effects of inhaled and orally ingested Delta-8 THC in comparison to both placebo and Delta-9 THC. Delta-8 THC is an cannabinoid that has become widely available for retail sale in the US due to a loophole in the 2018 Farm Bill. Delta-8 THC is an isomer of Delta-9 THC, which is the compound responsible for most of the psychoactive effects associated with cannabis. Prior research, while limited, has indicated that Delta-8 THC is less potent but has comparable pharmacodynamic effects to Delta-9 THC, especially at higher doses. The purpose of this study is to assess the effects of Delta-8 THC as compared to placebo and Delta-9 THC. Oral fluid, urine, blood, and hair specimens will be collected from participants. The investigators will recruit healthy participants between the ages of 18 and 45 who have prior experience using THC but have not used in at least one month. Two sub-studies will be run, with 5 conditions in each study; sub-study 1 will examine the effects of vaporized Delta-8 THC and sub-study 2 will assess the effects of orally ingested Delta-8 THC. Participants can complete both sub-studies but it is not required. There will be a minimum of 5 outpatient drug administration sessions for each participant, with the option to complete 5 more if interested. The investigators will recruit and consent up to 70 participants in order to obtain 20 completers (up to 40 total individuals) for each sub-study.

ELIGIBILITY:
Inclusion Criteria:

1. Have provided written informed consent
2. Be between the ages of 18 and 45
3. Be in good general health based on a physical examination, medical history, vital signs, and screening urine and blood tests
4. Test negative for recent cannabis use in urine at the screening visit and again upon admission for each experimental session
5. Test negative for other drugs of abuse, including alcohol at the screening visit and upon arrival for each experimental session
6. Not be pregnant or nursing (if female). All females must have a negative serum pregnancy test at the screening visit and a negative urine pregnancy test at clinic admission.
7. Have a body mass index (BMI) in the range of 19 to 36 kg/m2
8. Blood pressure at Screening Visit does not exceed a systolic blood pressure (SBP) of 150 mmHg or a diastolic blood pressure (DBP) of 90 mmHg
9. Report prior experience inhaling cannabis (either via smoking or vaporization).
10. Have not donated blood in the prior 30 days.

Exclusion Criteria:

1. Non-medical use of psychoactive drugs other than, nicotine, alcohol, or caffeine in the month prior to the Screening Visit;
2. History of or current evidence of significant medical or psychiatric illness judged by the investigator to put the participant at greater risk of experiencing an adverse event due to exposure or completion of other study procedures.
3. Use of an over-the-counter (OTC), systemic or topical drug(s), herbal supplement(s), or vitamin(s) within 14 days of experimental sessions; which, in the opinion of the investigator or sponsor, will interfere with the study result or the safety of the subject.
4. Use of a prescription medication (with the exception of birth control prescriptions) within 14 days of experimental sessions; which, in the opinion of the investigator or sponsor, will interfere with the study result or the safety of the subject. This includes any medication metabolized via CYP2D6, CYP2C9, CYP2B10, or which induce/inhibit CYP3A4 enzymes.
5. Use of any hemp, cannabis or cannabinoid product in the past 3 months.
6. History of xerostomia (dry mouth), or the presence of mucositis, gum infection or bleeding, or other significant oral cavity disease or disorder that in the investigator's opinion may affect the collection of oral fluid samples.
7. History of clinically significant cardiac arrhythmias or vasospastic disease (e.g., Prinzmetal's angina).
8. Enrolled in another clinical trial or have received any drug as part of a research study within 30 days prior to dosing.
9. Epilepsy or a history of seizures.
10. Individuals who have a recent history of traumatic brain injury diagnosed by CT/MRI and have current sequela from prior brain injury, as determined by the study physician.
11. Individuals with anemia judged by medical staff to place the person at risk due to the frequency and volume of blood collected during the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2024-08-08 (Actual); Study Completion 2024-10-02 (Actual)

PRIMARY OUTCOMES:
Self-reported Drug Effect ratings on the Drug Effect Questionnaire (DEQ) | Within 8 hours
  Subjective drug effect ratings (0-100) will be collected with the Drug Effect Questionnaire, with 0 being no effect and 100 being maximum effect.

SECONDARY OUTCOMES:
Behavioral task performance as assessed by the DRUID app | Within 8 hours
  Composite score on the DRUID App, a measure of behavioral task performance (range 0-100) where lower scores indicate better performance.
Quantitative levels of D-9-THC in blood | Within 8 hours
  Blood is collected through an intravenous catheter, quantitative results are reported in nanograms per milliliter (ng/ml).
Quantitative levels of D-8-THC in blood | Within 8 hours
  Blood is collected through an intravenous catheter, quantitative results are reported in nanograms per milliliter (ng/ml).
Paced Auditory Serial Addition Task (PASAT) score | Within 8 hours
  Paced Auditory Serial Addition Task, cognitive task that measures cognitive function by assessing auditory information processing speed and flexibility, as well as calculation ability.
Digit Symbol Substitution Task (DSST) score | Within 8 hours
  Digit Symbol Substitution Task, cognitive task administered to assess response speed, sustained attention, visual spatial skills and set shifting.
Divided Attention as assessed by the DAT | Within 8 hours
  Divided Attention Task (DAT), cognitive task administered on the computer to assess divided attention.
Heart rate | Within 8 hours
  Heart rate (beats/minute) will be measured while sitting down using the vitals machine.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Vandrey, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Behavioral Pharmacology Research Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No